CLINICAL TRIAL: NCT03508596
Title: STRAIN - Work-related Stress Among Health Professionals in Switzerland
Acronym: STRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sabine Hahn (Other)
Collaborators: University of Applied Sciences and Arts of Southern Switzerland (Other); University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Sponsor-Investigator, Sabine Hahn, Head of Nursing Division, Division Head of Applied Research & Development in Nursing, PhD, RN, Bern University of Applied Sciences
Organization: Bern University of Applied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: J.008137-42-PFLW
Record Dates: First submitted 2018-03-23; First posted 2018-04-26 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Stress; Health Care Professionals; Work-Related Condition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Intervention group (IG)
  An educational intervention for the supervisors
  Interventions: Other: educational intervention for the supervisors
- Control (No Intervention): control group (CG)
- Non-Intervention (No Intervention): group without intervention (GWI)

INTERVENTIONS:
Other: educational intervention for the supervisors — The educational intervention is based on a systematic literature review as well as focus-group interviews with health care professionals. It will be developed until the end of 2018
  Arms: Intervention

SUMMARY:
The aim of this study is to identify work stressors, stress reactions and long-term consequences among nurses, physicians, medical-technical and medical-therapeutic professions in Switzerland and to reduce those factors by an educational intervention for the supervisors.

DETAILED DESCRIPTION:
Methods: This study is a cross-sectional design and randomly selected hospitals, nursing homes and home care organizations. The study sample included nursing staff and midwives, physicians, medical-technical and medical-therapeutic professionals at all hierarchical levels. Data were collected using self-report questionnaires and analysed using multiple regression models.

ELIGIBILITY:
Inclusion Criteria:

* Employee within a participating health organization in Switzerland
* Health care professional (nurse, medical-technical medical-therapeutical profession, physician)

Exclusion Criteria:

* Health professionals without an fixed employment contract

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8112 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
effort reward imbalance model (ERI) | Changes in self reported results of the ERI from t1 to t2 (1 year)
  The model defines threatening job conditions as a "mismatch between high workload (high demand) and low control over long-term rewards"

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hahn, Study Director — Bern University of Applied Sciences Switzerland

IPD SHARING:
Plan to Share IPD: No